CLINICAL TRIAL: NCT04456933
Title: RESECTION AND INTRACORPOREAL ANASTOMOSIS IN LAPAROSCOPIC LEFT COLECTOMY AS AN ADAPTATION TO THE PANDEMIC CAUSED BY SARS-CoV-2 (COVID19). A COMPARATIVE COHORT STUDY
Brief Title: Intracorporeal Anastomosis in Laparoscopic Left Colectomy. Cohort Comparative Study
Acronym: RIAL-COLECTOMY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Irene Gómez Torres (Unknown); Laura Mora López (Unknown); Anna Pallisera-Lloveras (Unknown); Sheila Serra-Pla (Unknown); Albert García Nalda (Unknown); Anna Serracant-Barrera (Unknown); Mercedes Muñoz (Unknown); Oriol Pino-Pérez (Unknown)
Responsible Party: Principal Investigator, Xavier Serra-Aracil, Head of Colorectal Unit, Corporacion Parc Tauli
Other Study IDs: HEMI-E-INTRACORPOREA-2020
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Colon Cancer
Keywords: Left Colon Cancer,; Left hemicolectomy; Laparoscopic left hemicolectomy; Intracorporeal resection and anastomosis
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Extracorporeal left hemicolectomy anastomosis — Standard surgical technique protocolized in the unit for laparoscopic surgery of the left colon, sigma and high rectum for the last 10 years.
  After sectioning the distal colon using a mechanical stapler (60mm blue load), a pfannestiel-type suprapubic accessory incision is made, with externalization of the tumor under wound protection with a ringed retraction device. Both the resection of the left mesocolon or mesosigma, and the placement of the head of the circular stapler are performed extracorporeally by proximal section of the colon with a pursetring® self-suturing device, removal of the piece, placement of the head, and reconnection of the pneumoperitoneum for colorectal anastomosis with Circular Stapler Curved B. Braun®
Procedure: Intracorporeal left hemicolectomy anastomosis — o Intracorporeal resection of the left mesocolon
  The mesocolon resection will be performed totally intracorporeally to its proximal end. The distal colon section will be performed using a mechanical stapler (blue charge 60mm)
  o Preparation of Intracorporeal Anastomosis
  The anastomosis will be performed in a mechanical end-to-end manner using a Circular Stapler Curved B. Braun®.
  The Insertion of the stapler head into the proximal colon will be placed intracorporeally with an incision distal to the staple section. Once the head has been exteriorized at the terminal end of the proximal colon, a circular purse-type suture with prolene 2.0 will be made.
  Once the mechanical colorectal anastomosis is performed, 4-6 stitches of anastomotic reinforcement with silk 2.0 will be placed.
  The extraction of the piece will be carried out with endobag protection and with an accessory incision (pfannestiel or other location depending on the patient)

SUMMARY:
OBJECTIVE: The aim of the study is to demonstrate that the intracorporeal resection and anastomosis in left-sided colon cancer, sigma and upper rectum, is not inferior to extracoprporeal resection and anastomosis, in terms of anastomotic leakage.

BACKGROUND: Due to the recent events of a pandemic respiratory disease secondary to infection by SARS-CoV-2 virus or coronavirus 19 (COVID19), surgeons have been forced to adapt our surgical procedures in order to minimize exposure to the virus as much as possible.

Based on the recommendations in case of surgery in patients with highly contagious viral diseases, the latest studies suggest minimally invasive accesses to minimize the risk of contagion. One of the proposed measures is the performance of intracorporeal anastomoses. Therefore, given the extensive experience of our center in minimally invasive surgery and studies on the validation of intracorporeal anastomosis techniques in both laparoscopic surgery of the right colon and rectum (TaTME), and the study of advantages that they can provide to the patient, our intention is to apply it to surgery on the left colon, sigma and upper rectum. Our hypothesis is that exteriorization of the colon through an accessory incision increases the risk of tension at the mesocolon level, thus increasing the risk of vascular deficit at the level of the staple area and it may increase the rate of anastomotic leakage. In this sense, studies that validate a standard technique of intracorporeal anastomosis in left colon surgery and that demonstrate its benefit with respect to extracorporeal anastomosis are lacking. We intend to describe a new intracorporeal anastomosis technique (ICA) that is feasible and safe for the patient and that can be applied universally. Once the ICA technique is established, it will allow us to determine its non-inferiority compared to the standard technique performed up to now with extracorporeal anastomosis.

METHODS: All consecutive patients with left-sided, sigma and upper rectum adenocarcinoma will be included into a prospective cohort and treated by laparoscopy with totally intracorporeal resection and anastomosis. They will be compared with a retrospective cohort of consecutive patients of identical characteristics treated by laparoscopy with extracorporeal resection and anastomosis, in the immediate chronological period.

DETAILED DESCRIPTION:
HYPOTHESIS Resection of the left colon / sigmoid with intracorporeal colorectal TT anastomosis is safe and not inferior to that performed extracorporeally. With the benefits of reduced intraoperative dissection, traction on the mesenteries, reduced vascular compromise of the anastomosis, a smaller incision size and being able to choose its location.

Main Aim:

The objective of this study is to demonstrate that colorectal mechanical end-to-end intracorporeal anastomosis is not inferior to extracorporeal approach in terms of anastomotic dehiscence.

Secondary Aims:

* To demonstrate the reproducibility of the colorectal mechanical end-to-end intracorporeal anastomosis technique in terms of reconversion, anastomotic dehiscence, organo-cavitary infection, and other postoperative complications.
* To determine the benefits that the IC anastomosis technique can bring to patients with obesity.
* To determine the benefits that the IC anastomosis technique can provide in terms of postoperative complications, hospital stay, and size of the accessory incision.
* To determine the benefit of the application of indocyanine green to determine the point of resection and anastomosis.

STUDY DESIGN

Comparative, single-center, controlled non-inferiority cohort study of resection and mechanical end-to-end intracorporeal anastomosis in left colon, sigmoid, and upper rectum surgery (prospective cohort) versus the standard technique of extracorporeal laparoscopic surgery (retrospective cohort).

SUBJECTS OF THE STUDY

In group 1 or control (retrospective cohort): patients diagnosed with adenocarcinoma of the left colon, sigmoid or upper rectum who meet the inclusion criteria Operated on surgically by our unit, collected in our database, by laparoscopic oncological surgery applying the conventional extracorporeal anastomosis technique.

In group 2 or case (prospective cohort): patients diagnosed with adenocarcinoma of the left colon, sigmoid or upper rectum, that meet the inclusion criteria, with an oncological surgical indication with a laparoscopic approach since July 2020, to which the resection and intracoporeal anastomosis technique will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Left Colonic Adenocarcinoma. Location of the tumor in the left colon, sigma or high rectum (with the anastomosis performed above the peritoneal reflection). Non-metastatic stage. Scheduled oncological surgery with curative intention operated on with laparoscopic surgery with resection technique and intracorporeal anastomosis. Over 18 years

Exclusion Criteria:

* Other tumor locations. Non-adenocarcinoma tumors. Synchronous tumors. T4 tumor stage and stage IV of TNM classification. ASA IV (American Society of Anesthesiologists). Non-optimal nutritional study (preoperative albumin ≤3.4 g / dl). Do not sign informed consent. Pregnant patients. Diagnosis of another type of neoplasm with active disease. Liver cirrhosis, Chronic kidney failure on dialysis treatment, patients with stent bridge to elective surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In group 1 or control (retrospective cohort): patients diagnosed with adenocarcinoma of the left colon, sigmoid or upper rectum who meet the inclusion criteria Operated on surgically by our unit, collected in our database, by laparoscopic oncological surgery applying the conventional extracorporeal anastomosis technique.
  In group 2 or case (prospective cohort): patients diagnosed with adenocarcinoma of the left colon, sigmoid or upper rectum, that meet the inclusion criteria, with an oncological surgical indication with a laparoscopic approach since July 2020, to which the resection and intracoporeal anastomosis technique will be applied.
Sampling Method: Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of anastomotic leak (AL) | 30 days
  Percentage of anastomic leak (defined in accordance with Peel et al.).

SECONDARY OUTCOMES:
Rate of global morbidity | 30 days
  Dindo-Clavien Classification
Rate of Surgical site infection | 30 days
  SSI in accordance with the Center for Disease Control (CDC) National
Rate of Re-interventions | 30 days
  Percentage of re-interventions due to surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Serra-Aracil, MD,PhD, Principal Investigator — Corporacio Parc Tauli. Parc Tauli University Hospital
Locations (1):
- Hospital Universitario Parc Tauli de Sabadel, Sabadell, Barceelona, Spain

REFERENCES:
- [Background] Serra-Aracil X, Mora-Lopez L, Casalots A, Pericay C, Guerrero R, Navarro-Soto S. Hybrid NOTES: TEO for transanal total mesorectal excision: intracorporeal resection and anastomosis. Surg Endosc. 2016 Jan;30(1):346-54. doi: 10.1007/s00464-015-4170-5. Epub 2015 Mar 27. PMID 25814073
- [Background] Akamatsu H, Omori T, Oyama T, Tori M, Ueshima S, Nakahara M, Abe T, Nishida T. Totally laparoscopic sigmoid colectomy: a simple and safe technique for intracorporeal anastomosis. Surg Endosc. 2009 Nov;23(11):2605-9. doi: 10.1007/s00464-009-0406-6. Epub 2009 Mar 6. PMID 19266229